CLINICAL TRIAL: NCT04362878
Title: Evaluation of Mental Health, Self-esteem, Body Image and Quality of Life in Patients With Pectus Excavatum or Pectus Carinatum: Relationship With Severity and Type of the Deformity, and Patients' Age
Brief Title: Psychological Assessment of Patients With Chest Wall Deformities
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Daniela Graziani, Principal Investigator, University of Florence
Other Study IDs: 176/2019
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Pectus Excavatum; Pectus Carinatum
Keywords: Pectus excavatum; Pectus carinatum; Adolescents; Psychological Assessment; Quality of life
MeSH Terms: conditions — Funnel Chest; Pectus Carinatum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to investigate the most frequent psychological outcomes associated to chest wall deformities and patients' quality of life.

DETAILED DESCRIPTION:
The study aims at providing psychological assessment (body image, self-esteem, overall mental health) and quality of life investigation of adolescents affected by chest wall deformities, in relation to the severity and type of deformity, and patients' age; identifying risk factors for psychological disorders.

The following hypotheses were tested: differences between patients with different chest wall deformities regarding body image and mental health were expected; no hypothesis on the possible results concerning the effect of the severity of deformity on each studied variable was formulated, since previous findings are unclear. Concerning age, some differences according to different age ranges were expected. Regarding risk factors for mental health problems, older age and greater body image dissatisfaction were expected to be significant risk factors for psychological problems; regarding the severity and type of deformity, results of previous studies are unclear or lacking, so no hypothesis was tested; quality of life and self-esteem variables were also tested, as previous studies showed they are significantly related to general well being and mental health in adolescents.

Adolescents coming at the outpatient clinics for the first evaluation of their chest wall and one of their parents/caregivers were enrolled. After the medical examination, patients meeting inclusion criteria are invited to participate in the study and to be assessed by a trained psychologist who administered them all questionnaires after they expressed their informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pectus excavatum or pectus carinatum;
* Age from 12 to 18 years old;
* High level of fluency in Italian.

Exclusion Criteria:

* Clinical diagnosis of chronic or acute disease, or presence of other conditions which could significantly influence adolescents' quality of life, mental health, body image and self-esteem;
* Diagnosis of intellectual disability or other conditions (e.g. low level of fluency in Italian) which could hinder questionnaires understanding.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents coming for the first medical examination of their chest wall at the Pectus Center outpatient clinic will be invited to participate in the study. Adolescents who express their voluntary participation will be enrolled. One of their parents/caregivers is also invited to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Differences in mental health mean scores on the Youth Self-Report (YSR) among patients with different severity indexes. | Baseline.
  The YSR 11-18 is a validated self-report measure of 11-18 years old adolescents' social competences, behavioral and emotional problems. Different cut-off scores are provided according to age and gender to identify scores in the normal, borderline or clinical range.
Differences in mental health mean scores on the Youth Self-Report (YSR) between PE and PC patients. | Baseline
  The YSR 11-18 is a validated self-report measure of 11-18 years old adolescents' social competences, behavioral and emotional problems. Different cut-off scores are provided according to age and gender to identify scores in the normal, borderline or clinical range.
Differences in mental health mean scores on the Youth Self-Report (YSR) among patients in different age ranges. | Baseline
  The YSR 11-18 is a validated self-report measure of 11-18 years old adolescents' social competences, behavioral and emotional problems. Different cut-off scores are provided according to age and gender to identify scores in the normal, borderline or clinical range.
Correlation between mental health scores on the Child Behavior Checklist (CBCL) and mental health scores on the Youth Self-Report (YSR). | Baseline.
  The CBCL 6-18 is a questionnaire to be filled out by parents to assess social competence and behavioral and emotional problems in children and adolescents aged 6 to 18 years old; different cut-off scores are provided according to children's/adolescents' age and gender to identify scores in the normal, borderline or clinical range.

SECONDARY OUTCOMES:
Differences in body image mean scores on the Body Uneasiness Test (BUT) among patients with different severity indexes. | Baseline.
  The BUT is a self-report measure of the overall body perception (BUT-A) and specific body parts or functions perception (BUT-B). It has been validated on a sample of participants from 13 to over 65 years old. Higher scores correspond to greater body uneasiness.
Differences in body image mean scores on the Body Uneasiness Test (BUT) between PE and PC patients. | Baseline.
  The BUT is a self-report measure of the overall body perception (BUT-A) and specific body parts or functions perception (BUT-B). It has been validated on a sample of participants from 13 to over 65 years old. Higher scores correspond to greater body uneasiness.
Differences in body image mean scores on the Body Uneasiness Test (BUT) among patients in different age ranges. | Baseline.
  The BUT is a self-report measure of the overall body perception (BUT-A) and specific body parts or functions perception (BUT-B). It has been validated on a sample of participants from 13 to over 65 years old. Higher scores correspond to greater body uneasiness.
Correlation among body image scores on the Body Uneasiness Test (BUT) and mental health scores on the Youth Self-Report (YSR). | Baseline.
  The BUT is a self-report measure of the overall body perception (BUT-A) and specific body parts or functions perception (BUT-B). It has been validated on a sample of participants from 13 to over 65 years old. Higher scores correspond to greater body uneasiness.
Differences in self-esteem mean scores on the Rosenberg Self-Esteem Scale (RSES) among patients with different severity indexes. | Baseline.
  The RSES is validated self-report measures of self-esteem, widely used in adolescents. Higher scores correspond to higher self-esteem. A score of lower than 15 indicates low self-esteem.
Differences in self-esteem mean scores on the Rosenberg Self-Esteem Scale (RSES) between PE and PC patients. | Baseline.
  The RSES is validated self-report measures of self-esteem, widely used in adolescents. Higher scores correspond to higher self-esteem. A score of lower than 15 indicates low self-esteem.
Differences in self-esteem mean scores on the Rosenberg Self-Esteem Scale (RSES) among patients in different age ranges. | Baseline.
  The RSES is validated self-report measures of self-esteem, widely used in adolescents. Higher scores correspond to higher self-esteem. A score of lower than 15 indicates low self-esteem.
Correlation among self-esteem scores on the Rosenberg Self-Esteem Scale (RSES) and mental health scores on the Youth Self-Report (YSR). | Baseline.
  The RSES is validated self-report measures of self-esteem, widely used in adolescents. Higher scores correspond to higher self-esteem. A score of lower than 15 indicates low self-esteem.
Differences in quality of life mean scores on the Pediatric Quality of life Inventory (Peds-Ql) among patients with different severity indexes. | Baseline.
  The Peds-Ql is a validated self-report measure of the quality of life in children and adolescents in different age ranges. For the present study, the 8-12 years old early-adolescents version and the 13-18 years old adolescents version are used. Higher scores indicated a better quality of life.
Differences in quality of life mean scores on the Pediatric Quality of life Inventory (Peds-Ql) between PE and PC patients. | Baseline.
  The Peds-Ql is a validated self-report measure of the quality of life in children and adolescents in different age ranges. For the present study, the 8-12 years old early-adolescents version and the 13-18 years old adolescents version are used. Higher scores indicated a better quality of life.
Differences in quality of life mean scores on the Pediatric Quality of life Inventory (Peds-Ql) among patients in different age ranges. | Baseline.
  The Peds-Ql is a validated self-report measure of the quality of life in children and adolescents in different age ranges. For the present study, the 8-12 years old early-adolescents version and the 13-18 years old adolescents version are used. Higher scores indicated a better quality of life.
Correlation among quality of life scores on the Pediatric Quality of life Inventory (Peds-Ql) and mental health scores on the Youth Self-Report (YSR). | Baseline.
  The Peds-Ql is a validated self-report measure of the quality of life in children and adolescents in different age ranges. For the present study, the 8-12 years old early-adolescents version and the 13-18 years old adolescents version are used. Higher scores indicated a better quality of life.
Correlation between scores on Pediatric Quality of Life Inventory (parent version) and scores on Pediatric Quality of Life Inventory (early-adolescent and adolescent versions). | One only time point, immediately after the medical examination, that requires 10 minutes for questionnaire completion.
  The Peds-Ql (parent version) is a validated tool filled out by parents of children and adolescents in different age ranges. For the present study, the 8-12 years old early-adolescents' parent version and the 13-18 years old adolescents' parent version are used. Higher scores indicated a better quality of life.

OTHER OUTCOMES:
Degree of the severity of malformation rated on a six-point classification. | Baseline.
  The severity of the deformity was rated according to six severity classes, from 0= absent to 5=extremely severe. This classification method was developed from a 3D scanner procedure and it demonstrated to outperform traditional classification methods.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rosanna, PsyD, Study Director — Meyer Children's Hospital IRCCS
Locations (1):
- Meyer Children's Hospital, Florence, Italy

REFERENCES:
- [Background] Li H, Jin X, Fan S, Wang D, Wu C, Pan Z, Li Y, An Y, Wang G, Dai J, Wang Q. Behavioural disorders in children with pectus excavatum in China: a retrospective cohort study with propensity score matching and risk prediction model. Eur J Cardiothorac Surg. 2019 Sep 1;56(3):596-603. doi: 10.1093/ejcts/ezz038. PMID 30824916
- [Background] Steinmann C, Krille S, Mueller A, Weber P, Reingruber B, Martin A. Pectus excavatum and pectus carinatum patients suffer from lower quality of life and impaired body image: a control group comparison of psychological characteristics prior to surgical correction. Eur J Cardiothorac Surg. 2011 Nov;40(5):1138-45. doi: 10.1016/j.ejcts.2011.02.019. Epub 2011 Mar 25. PMID 21440452
- [Background] Luo L, Xu B, Wang X, Tan B, Zhao J. Intervention of the Nuss Procedure on the Mental Health of Pectus Excavatum Patients. Ann Thorac Cardiovasc Surg. 2017 Aug 20;23(4):175-180. doi: 10.5761/atcs.oa.17-00014. Epub 2017 Jun 16. PMID 28626162
- [Background] Hadolt B, Wallisch A, Egger JW, Hollwarth ME. Body-image, self-concept and mental exposure in patients with pectus excavatum. Pediatr Surg Int. 2011 Jun;27(6):665-70. doi: 10.1007/s00383-011-2854-z. Epub 2011 Feb 3. PMID 21290134
- [Background] Ji Y, Liu W, Chen S, Xu B, Tang Y, Wang X, Yang G, Cao L. Assessment of psychosocial functioning and its risk factors in children with pectus excavatum. Health Qual Life Outcomes. 2011 May 4;9:28. doi: 10.1186/1477-7525-9-28. PMID 21542911
- [Background] Ticchi D, Eisinger RS, Pilegaard HK, Torre M, Sesia SB, Infante M, Voulaz E, Quesada MA, Sisask M. Evaluating interest in narrative therapy for decision making about pectus excavatum treatment. Interact Cardiovasc Thorac Surg. 2018 Feb 1;26(2):271-275. doi: 10.1093/icvts/ivx308. PMID 29049840
- [Background] Wildemeersch D, Bernaerts L, D'Hondt M, Hans G. Reference Correction: Preliminary Evaluation of a Web-Based Psychological Screening Tool in Adolescents Undergoing Minimally Invasive Pectus Surgery: Single-Center Observational Cohort Study. JMIR Ment Health. 2018 Nov 12;5(4):e11608. doi: 10.2196/11608. PMID 30578210